CLINICAL TRIAL: NCT05898204
Title: Comparison of the Effects of a Ketogenic Diet and an Isocaloric Balanced Diet in Obese Patients: a Randomized Clinical Trial
Brief Title: KEtogenic Diet and Its Multiple EffectS on Obesity
Acronym: KEMESO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lucio Gnessi, Full Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEMESO1
Record Dates: First submitted 2023-04-25; First posted 2023-06-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: obesity; metabolism; circadian rhythm; sleep; quality of life; balanced diet; ketogenic diet; immune profile
MeSH Terms: conditions — Obesity | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Patients are sequentially allocated to one of the 2 arms of intervention: the ketogenic diet arm or the balanced diet arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketogenic diet arm (Experimental): Ketogenic diet for a month, or a longer period if clinically necessary
  Interventions: Other: Ketogenic diet
- Balanced diet arm (Active Comparator): Balanced diet for a month, or a longer period if clinically necessary
  Interventions: Other: Balanced diet

INTERVENTIONS:
Other: Ketogenic diet — Prescription of a ketogenic diet, 1200 Kcal/die. Patients are encouraged to walk 30 minutes every day.
  Arms: Ketogenic diet arm
Other: Balanced diet — Prescription of a balanced diet, 1200 Kcal/die. Patients are encouraged to walk 30 minutes every day.
  Arms: Balanced diet arm

SUMMARY:
The prevalence of obesity and metabolic disturbances is worryingly increasing worldwide, therefore the study of their pathophysiology is extremely important to find new strategies for their treatment. Obesity has a strong impact not only on the metabolism of the patients, but also may impact hormonal, inflammatory and immune profile, and profoundly influence the daily life of the patients. Weight loss may determine an amelioration of these parameters, but the impact of the diet composition aimed to weight loss on them has not been profoundly studied yet.

The aim of our research project is to study the effects of a ketogenic diet in comparison with an isocaloric balanced diet on weight loss and anthropometric parameters, quality of life, hormone profile, sleep, sexual function, circadian rhythm, inflammatory and immunological parameters in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* BMI≥ 30 Kg/m2

Exclusion Criteria:

* Type 1 diabetes mellitus and latent autoimmune diabetes in adults
* β-cell failure in type 2 diabetes mellitus
* Use of sodium/glucose cotransporter 2 (SGLT2) inhibitors
* Pregnancy and breastfeeding
* Kidney failure and moderate-to-severe chronic kidney disease
* Liver failure
* Heart failure (NYHA III-IV)
* Respiratory failure
* Unstable angina, stroke or myocardial infarction in the last 12 months
* Cardiac arrhythmias
* Eating disorders and other severe mental illnesses, alcohol and substance abuse
* Active/severe infections
* Planned elective surgery or invasive procedures
* Rare disorders: porphyria, carnitine deficiency, carnitine palmitoyltransferase deficiency, carnitine-acylcarnitine translocase deficiency, mitochondrial fatty acid β-oxidation disorders, pyruvate carboxylase deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of changes in Perceived Quality of Life with IWQOL-Lite Questionnaires | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessment with the questionnaires Impact of weight/Quality of Life-Lite (IWQOL-Lite); global scale from 0 to 100; the higher the score, the better the quality of life
Evaluation of changes in Perceived Quality of Life with SF-36 Questionnaires | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessment with the questionnaires Short Form Health Survey 36 (SF-36); scale of every item from 0 to 100; the higher the score, the better the quality of life
Evaluation of changes in Perceived Quality of Life with "EQ-5D" Questionnaires | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessment with the questionnaires "EQ-5D"; scale of every item from 1 to 5; the higher the score, the worse the perceived problem

SECONDARY OUTCOMES:
Evaluation of weight loss | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Weight loss expressed in Kg
Evaluation of changes of perceived sleep | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessment with the questionnaires Pittsburgh Sleep Quality Index; global score on a scale from 0 to 21; the higher the score, the worse the sleep quality
Evaluation of changes of perceived sleepiness | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessment with the questionnaires Epworth Sleepiness Scale (ESS); score on a scale from 0 to 24; the higher the score, the higher the sleepiness
Evaluation of changes in clock genes expression | At baseline, at 30 days
  Evaluation of the expression of the clock genes in blood cells
Evaluation of changes in hormonal profile | At baseline, at 30 days
  Assessment of hormonal parameters, as cortisol, expressed in ug/dL
Evaluation of changes in sexual function in males | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessed with the questionnaires International Index of Erectile Function (IIEF-5); scale from 5 to 25; the higher the score, the better the erectile function
Evaluation of changes in inflammation | At baseline, at 30 days, at 60 days if the patient continued the diet
  Measurements of circulating cytokines, as interleukin 2 and interleukin 10, expressed in ng/mL
Evaluation of changes of peripheral blood mononuclear cells | At baseline, at 30 days, at 60 days if the patient continued the diet
  Number of cells of peripheral blood mononuclear cell subpopulations, expressed in number/mm3
Evaluation of changes in sleep parameters (length) | At baseline, at 30 days
  Assessment with actigraphy of latency, total minutes in bed, total sleep time, wake after sleep onset, average awakening length, expressed in minutes
Evaluation of changes in hip circumference | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessment of hip circumference, expressed in cm
Evaluation of changes in waist circumference | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessment of waist circumference, expressed in cm
Change in circadian rhythm | At baseline, at 30 days
  Evaluation of change in midpoint of sleep, bedtime, sleep onset, rise time and circadian phase, expressed in hours
Evaluation of changes in Sexual Function in Females | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Assessed with the questionnaire Female Sexual Function Index (FSFI); scale of every item from 1 to 5; the higher score, the better the sexual function
Evaluation of changes in sleep efficiency | At baseline, at 30 days
  Sleep efficiency expressed as a percentage; measurement with actigraphy
Evaluation of changes in number of awakenings | At baseline, at 30 days
  Measurement with actigraphy
Evaluation of changes in sleep parameters | At baseline, at 30 days
  Evaluation of sleep fragmentation index and movement index, with actigraphy
Evaluation of changes in metabolic parameters | At baseline, at 30 days
  Evaluation of changes in metabolic parameters, as glucose, triglycerides, cholesterol and HDL, expressed in mmol/L
Evaluation of changes in BMI | At baseline, at 15 days, at 30 days, at 60 days if the patient continued the diet
  Weight and height will be combined to report BMI in kg/m^2
Evaluation of height | At baseline
  Assessment of height, expressed in cm
Evaluation of changes in whole blood cells gene expression | At baseline, at 30 days
  Evaluation of the changes in the expression of blood cells genes, as metabolic, inflammatory and immunological genes, with RNA-seq in whole blood cells

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No